CLINICAL TRIAL: NCT05477901
Title: Mental Health and Bolsa Familia: A Mechanistically Focused Clinical Trial of a Cash Transfer Intervention on Child Brain, Behavior, and Mental Health
Brief Title: Impacts of Cash Transfers on Child Neurodevelopment (Auxilio Brasil)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cristiane Duarte, Ruane Professor for the Implementation of Science for Child and Adolescent mental Health (in Psychiatry) at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #8245; 1R01MH128937-01 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-07-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Inflammation; HPA; CBCL; Family Relations
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Post-baseline Procedure -- Random Assignment to Intervention After baseline, families will be randomized in a 1:1 ratio to receive either a high ($40/month) or low ($2/month) supplemental transfer for 2 years and remains in their study arm throughout the study after randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): High supplemental transfer: $40 a month
  Interventions: Other: Supplemental cash transfer
- Control (No Intervention): Low supplemental transfer: $2 a month

INTERVENTIONS:
Other: Supplemental cash transfer — Supplemental cash transfer ($40/month)
  Arms: Intervention

SUMMARY:
This study examines the impact of Auxilio Brasil (AB), a cash transfer program to mothers of school-age children, on resource-deprived populations in Brazil and its protective effects on child neurodevelopment and mental health. The investigators will conduct a randomized clinical trial (RCT) among those already receiving AB in which 300 families will be randomized in a 1:1 ratio to receive either a high ($40/month) or low ($2/month) supplemental transfer for 2 years. Three hundred children (index child participants; 7-10 years old) will be enrolled across both study arms. Additionally, up to 150 siblings ("sibling participants;" 7-10 years old) will be enrolled. Eligible families who decide to participate will sign a study-specific informed consent (mother) and assent (child) form. The UNIFESP team will conduct the respective assessments at baseline, approximately 8- and 16- months, 24-months and approximately 6-months post-RCT.

Aim 1: Determine the impact of high vs low cash transfers on children's exposure to adversities (ACEs) and neurodevelopment.

Aim 2: Determine the impact of cash transfers on children's inflammatory markers and HPA activity/cortisol.

Exploratory Aim: The investigators will explore (i) whether sex/gender of the children moderates the pathways in the above mediation model; and (ii) whether cash transfer-related effects persist 6 months post-RCT.

DETAILED DESCRIPTION:
Numerous studies link childhood poverty with altered neurodevelopment with the most robust effects often in brain substrates related to executive functions (EF). Poverty is associated with reduced grey matter thickness and surface area of the prefrontal cortex (PFC), a key structure underlying EF (4,5) Poverty is also associated with altered structure and function of the hippocampus - a region essential for memory and cognitive control (5,6). Effects of poverty on brain development are thought to give rise to the well described associations between poverty, impairments in EF, and risk for mental illness (18). The possibility of lifting children out of poverty and thereby tempering poverty's malignant neurodevelopmental effects remains largely untested, particularly with brain and behavioral measures and within LMICs where poverty is widespread. To address this gap, the investigators propose a randomized clinical trial (RCT) to be conducted in low-income families in Sao Paulo, Brazil that will examine causal effects of a cash transfer program on neurodevelopment in youth. Our study builds off an existing cash transfer program (CTP) - Auxilio Brasil (AB) - and augments the cash transfer amount to a level sufficient to lift a family out of extreme poverty and poverty. Our RCT design will allow for novel causal inferences linking cash transfers to brain/behavior outcomes, while testing mechanistic hypotheses. Because the investigators are building off AB, a well-established program with a successful, national infrastructure for transferring cash, our findings could rapidly move toward implementation. Our study will inform critical unanswered questions about pasting, and CTPs generally, that could support their broader and more targeted implementation - First, if augmenting AB removes a family from poverty, does this protect child neurodevelopment? And second, if this augmented AB program protects neurodevelopment, what are the mechanisms that explain this? Providing this mechanistic framework is a key step toward refining AB and other CTPs, facilitating for example, studies aimed at targeting populations most likely to benefit, optimizing the dose/amount of the transfers, and determining the ideal timing/duration of CTPs.

Aims and Hypotheses

Aim 1: Determine the impact of high vs low cash transfers on children's exposure to adversities (ACEs) and neurodevelopment. Eligible families will be those already enrolled in Brazil's national AB program. Relative to low cash transfers, children of mothers who received high cash transfers will have:

Hypothesis 1A (H1A) - [ACEs] fewer new onset ACEs over the 24-month course of the RCT; H1B - [Neurodevelopment] greater pre-vs-post RCT increases in prefrontal activation during an EF fMRI task (Simon task),10 increased connectivity within EF-related PFC/mesolimbic circuits (resting fMRI and diffusion MRI), and improvements in EF behaviors.

Aim 2: Determine the impact of cash transfers on children's inflammatory markers and HPA activity/cortisol.

Hypothesis 2A (H2A) - Relative to low cash transfers, children of mothers who received high cash transfers will have lower pre vs-post RCT levels of pro-inflammatory markers (e.g., CRP, Il-6, TNF-a; from blood draws) and hair cortisol (HPA activity over past 2-3 months).

Hypothesis 2B (H2B) - Inflammatory and HPA activity levels (H2A) will be lower in children with fewer new onset ACEs (i.e., new ACEs occurring during the 24-month RCT). H2C [Mediation] - The effects of high cash transfers on neurodevelopment (H1B) will be mediated by the impact of cash transfers on reducing new onset ACEs (H1A) and lower inflammation and HPA activity (H2A & H2B), while taking into account covariates and three additional pathways (see A.9 And C.6.3).

Exploratory Aim: The investigators will explore (i) whether sex/gender of the children moderates the pathways in the above mediation model (H2C); and (ii) whether cash transfer-related effects - reducing new onset ACEs and symptoms (CBCL), and improved EF behavior - persist 6 months post-RCT.

Impact: Designed to decrease inequalities, AB is one of the largest social interventions in the world, yet its impact on child mental health is unknown. Our strategy, rather than relying on prohibitively expensive multi-site designs, proposes to generate evidence about the impact of AB on child neurodevelopmental outcomes by focusing on specific, well-supported mechanisms that may underlie mental illness risk. Our findings will have strong implications for tailoring the impact of cash transfer policies to maximize child mental health gains.

ELIGIBILITY:
Mother:

Inclusion Criteria:

1. Age 23-45 years old
2. Receiving AB cash transfers
3. Has at least two or more children ages 7- 10 years old at time of recruitment (up to 4 children per family)
4. Able to consent

Exclusion Criteria:

1. Mother and child do not reside in same household

Child:

Inclusion Criterion

1. Age 7-10 years old
2. Intellectual Disability

Exclusion Criterion

1. Does not reside in same household as the mother
2. Major Axis I disorder (e.g., Autism, Schizophrenia, Bipolar)
3. Severe Disability
4. MRI contradictions (index child only)

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Childhood Experiences (ACEs) - FHE | Baseline
  Family History Epidemiologic screener is a 9-item (+subitems) checklist to asses child's ACEs, more checked items mean more ACEs.
Changes in Adverse Childhood Experiences (ACEs) - FHE | 8 months
  Family History Epidemiologic screener is a 9-item (+subitems) checklist to asses child's ACEs, more checked items mean more ACEs.
Changes in Adverse Childhood Experiences (ACEs) - FHE | 16 months
  Family History Epidemiologic screener is a 9-item (+subitems) checklist to asses child's ACEs, more checked items mean more ACEs.
Changes in Adverse Childhood Experiences (ACEs) - FHE | 24 months
  Family History Epidemiologic screener is a 9-item (+subitems) checklist to asses child's ACEs, more checked items mean more ACEs.
Changes in Adverse Childhood Experiences (ACEs) - FHE | 6 months post-RCT
  Family History Epidemiologic screener is a 9-item (+subitems) checklist to asses child's ACEs, more checked items mean more ACEs.
Adverse Childhood Experiences (ACEs) - CTC | Baseline
  Brazilian version of the Parent-Child Conflict Tactics Scale: 22-item checklist with following subscales: non-violent discipline (NVD), psychological aggression (PSY), corporal punishment (CP), and physical maltreatment (PM). More checks in each subscales means behavior is performed more often.
Changes in Adverse Childhood Experiences (ACEs) - CTC | 8 months
  Brazilian version of the Parent-Child Conflict Tactics Scale: 22-item checklist with following subscales: non-violent discipline (NVD), psychological aggression (PSY), corporal punishment (CP), and physical maltreatment (PM). More checks in each subscales means behavior is performed more often.
Changes in Adverse Childhood Experiences (ACEs) - CTC | 16 months
  Brazilian version of the Parent-Child Conflict Tactics Scale: 22-item checklist with following subscales: non-violent discipline (NVD), psychological aggression (PSY), corporal punishment (CP), and physical maltreatment (PM). More checks in each subscales means behavior is performed more often.
Changes in Adverse Childhood Experiences (ACEs) - CTC | 24 months
  Brazilian version of the Parent-Child Conflict Tactics Scale: 22-item checklist with following subscales: non-violent discipline (NVD), psychological aggression (PSY), corporal punishment (CP), and physical maltreatment (PM). More checks in each subscales means behavior is performed more often.
Changes in Adverse Childhood Experiences (ACEs) - CTC | 6 months-post RCT
  Brazilian version of the Parent-Child Conflict Tactics Scale: 22-item checklist with following subscales: non-violent discipline (NVD), psychological aggression (PSY), corporal punishment (CP), and physical maltreatment (PM). More checks in each subscales means behavior is performed more often.
Child internalizing and externalizing symptoms | Baseline
  Maternal report of The Child Behavior Checklist, internalizing (score ranges from 0 to 33) and externalizing (score ranges from 0 to 35) scales. More checks in each scale means more internalizing or externalizing symptoms.
Changes in Child internalizing and externalizing symptoms | 8 months
  Maternal report of The Child Behavior Checklist, internalizing (score ranges from 0 to 33) and externalizing (score ranges from 0 to 35) scales. More checks in each scale mean more internalizing or externalizing symptoms.
Changes in Child internalizing and externalizing symptoms | 16 months
  Maternal report of The Child Behavior Checklist, internalizing (score ranges from 0 to 33) and externalizing (score ranges from 0 to 35) scales. More checks in each scale mean more internalizing or externalizing symptoms.
Changes in Child internalizing and externalizing symptoms | 24 months
  Maternal report of The Child Behavior Checklist, internalizing (score ranges from 0 to 33) and externalizing (score ranges from 0 to 35) scales. More checks in each scale mean more internalizing or externalizing symptoms.
Changes in Child internalizing and externalizing symptoms | 6 months-post RCT
  Maternal report of The Child Behavior Checklist, internalizing (score ranges from 0 to 33) and externalizing (score ranges from 0 to 35) scales. More checks in each scale mean more internalizing or externalizing symptoms.
Access to health care | Baseline
  The assessment will be based on maternal report about each child's health care utilization history including primary care, urgent care, and hospital care. Primary care visits will be classified by purpose: vaccination, routine check-up, or sick visits. Similar procedures to the ones in place in our ongoing study will be used to obtain child medical records in the primary care unit.
Changes in Access to health care | 8 months
  The assessment will be based on maternal report about each child's health care utilization history including primary care, urgent care, and hospital care. Primary care visits will be classified by purpose: vaccination, routine check-up, or sick visits. Similar procedures to the ones in place in our ongoing study will be used to obtain child medical records in the primary care unit.
Changes in Access to health care | 16 months
  The assessment will be based on maternal report about each child's health care utilization history including primary care, urgent care, and hospital care. Primary care visits will be classified by purpose: vaccination, routine check-up, or sick visits. Similar procedures to the ones in place in our ongoing study will be used to obtain child medical records in the primary care unit.
Changes in Access to health care | 24 months
  The assessment will be based on maternal report about each child's health care utilization history including primary care, urgent care, and hospital care. Primary care visits will be classified by purpose: vaccination, routine check-up, or sick visits. Similar procedures to the ones in place in our ongoing study will be used to obtain child medical records in the primary care unit.
Child brain MRI scan | Baseline
  Child participants will undergo an MRI scan (~1 hour) to examine the function and connectivity of EF-related brain systems
Changes in Child brain MRI scan | 24 months
  Child participants will undergo an MRI scan (~1 hour) to examine the function and connectivity of EF-related brain systems
Child Executive Function | Baseline
  Brazilian version of the Child Executive Functions Battery (CEF-B) assesses working memory, inhibition, flexibility and planning. Score ranges vary by domain. Higher scores mean higher capacity on specific domain.
Changes in Child Executive Function | 24 months
  Brazilian version of the Child Executive Functions Battery (CEF-B) assesses working memory, inhibition, flexibility and planning. Score ranges vary by domain. Higher scores mean higher capacity on specific domain.
Changes in Child Executive Function | 6 months-post RCT
  Brazilian version of the Child Executive Functions Battery (CEF-B) assesses working memory, inhibition, flexibility and planning. Score ranges vary by domain. Higher scores mean higher capacity on specific domain.
Biospecimen - Child hair sample | Baseline
  Child hair samples to measure HPA activity (cortisol)
Biospecimen - Changes in Child hair sample | 24 months
  Child hair samples to measure HPA activity(cortisol)
Biospecimen - Blood Draw - IL-6 | Baseline
  Primary immune measures will consist of IL-6 and CRP, consistent with prior research on inflammation and neurodevelopment.
Biospecimen - Blood Draw - Change in IL-6 | 24 months
  Primary immune measures will consist of IL-6 and CRP, consistent with prior research on inflammation and neurodevelopment.
Biospecimen - Blood Draw - CRP | Baseline
  Primary immune measures will consist of IL-6 and CRP, consistent with prior research on inflammation and neurodevelopment.
Biospecimen - Blood Draw - Change in CRP | 24 months
  Primary immune measures will consist of IL-6 and CRP, consistent with prior research on inflammation and neurodevelopment.
Family Adaptability and Cohesion Evaluation Scale-III (FACES-III) | Baseline
  This 20-item parent-report scale assesses family cohesion and adaptability. Cohesion: scores range from 0-50, higher scores mean a more cohesive family. Adaptability: scores range from 0-50, higher scores mean a more adaptable family.
Change in Family Adaptability and Cohesion Evaluation Scale-III (FACES-III) | 24 months
  This 20-item parent-report scale assesses family cohesion and adaptability. Cohesion: scores range from 0-50, higher scores mean a more cohesive family. Adaptability: scores range from 0-50, higher scores mean a more adaptable family.

SECONDARY OUTCOMES:
Food insecurity | Baseline, 24 months
  Mothers will be interviewed using the Brazilian adaptation of the Household Food insecurity. Scores range from 0-8. Higher scores mean more food insecurity.
Changes in Food insecurity | 24 months
  Mothers will be interviewed using the Brazilian adaptation of the Household Food insecurity. Scores range from 0-8. Higher scores mean more food insecurity.
Home observation/environment | Baseline
  The quality of the child's home environment will be assessed with the Home Observation Measurement of the Environment (HOME) Inventory. Scores range from 0 to 55. Higher scores mean more quality and quantity of stimulation and support available to child in the home.
Changes in Home observation/environment | 24 months
  The quality of the child's home environment will be assessed with the Home Observation Measurement of the Environment (HOME) Inventory. Scores range from 0 to 55. Higher scores mean more quality and quantity of stimulation and support available to child in the home.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Duarte, PhD, Principal Investigator — New York State Psychiatric Institute; Andrea Jackowsi, PhD, Principal Investigator — Federal University of São Paulo; Jonathan Posner, MD, Principal Investigator — Duke University; Tenneill Murray, MPH, Study Director — New York State Psychiatric Institute
Locations (2):
- New York State Psychiatric Institute, New York, New York, United States
- UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No